CLINICAL TRIAL: NCT03345966
Title: Validation of Assessment of Bmi-1 on Protein and Molecular Levels in Oral Dysplasia and Squamous Cell Carcinoma: A Diagnostic Study
Brief Title: Assessment of Bmi-1 on Protein and Molecular Levels in Oral Dysplasia and Squamous Cell Carcinoma: A Diagnostic Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Abo Gabal, teaching assistant, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CEBD-CU-2017-11-01
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Bmi-1 antibody using immunohistochemistry and PCR
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunohistochemistry (Experimental): In order to provide more precised data on Bmi-1 immunoexpression in OSCC, image analyzer will be used.
  The data will be obtained using the software (SIS, Germany), which comprise a light microscope (Olympus B × 60 Japan) capable of performing high speed digital image processing for the purpose of cell measurements. It will be calibrated automatically to convert the measurement units (pixels) produced by image analyzer program into actual micrometer units.
  Interventions: Diagnostic Test: Bmi-1 antibody
- Polymerase Chain Reaction PCR (Experimental): Calculation of Relative Quantification (RQ) (relative expression):
  After the RT-PCR will run, the data will be expressed in Cycle threshold (Ct).PCR data sheets will include Ct values of assessed gene and the house keeping (reference) gene which will be continuously expressed in the cell- (β-actin).To measure the gene expression of certain gene, -ve control sample shall be used. So target gene expression will be assessed and related to reference (internal control) gene as follows:
  Finally, RQ was calculated according to the following equation:
  1. ∆ Ct (Cycle threshold) = Ct assessed gene - Ct reference gene
  2. ∆∆ Ct = ∆ Ct sample - Ct control gene
  3. RQ = 2-(∆∆Ct)
  Interventions: Diagnostic Test: Bmi-1 antibody

INTERVENTIONS:
Diagnostic Test: Bmi-1 antibody — B-lymphoma Moloney murine leukemia virus insertion region-1
  Other Names: Expression of Bmi-1 molecule at RNA level by PCR and protein level by immunohistochemistry in oral dysplasia and squamous cell carcinoma

SUMMARY:
The aim of the current study is to assess the validation of Bmi-1 detection at both protein and molecular levels in oral epithelial dysplasia and oral squamous cell carcinoma as a biomarker for early cancer detection versus biopsy embedded in paraffin blocks.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) including oral squamous cell carcinoma (OSCC) has been reported as the sixth most common cause of cancer mortality in the world and the fifth most commonly occurring cancer. Thus a compelling need for investigation of the underlying molecular events associated with OSCC tumorigenesis has emerged for better understanding of such lesion. Moreover, identification of biomarkers for early detection and prediction of prognosis became of extreme importance, as it was reported that early diagnosis has been vital for effective treatment of OSCC and improved the survival rate of OSCC patients.

OSCC may originate from malignant transformation of the normal oral mucosa, as well as from oral potentially malignant lesions (OPMLs) with different degrees of oral epithelial dysplasia (OED). The approach of a step-wise transition from OPMLs to OSCC was well-established, but it could be difficult to predict if and when an OPML would undergo full transformation and resulted in a tumor. Thus, using specific molecular biomarkers able to identify OED lesions with higher potential for malignant transformation would be very beneficial. Unfortunately, up to date there has been no tools available to monitor OED lesions or HNSCC patients for early stages of local recurrences or distant metastases .

Among the recently introduced biomarkers, B-lymphoma Moloney murine leukemia virus insertion region-1 (BMI1), a member of the polycomb group (PcG) genes, was considered to be pivotal in regulating stemness-related genes involved in maintaining the self-renewal ability of stem cells by promoting chromatin modifications. BMI1 was also known to be deregulated in various human types of cancer. Previous studies have revealed the capability of BMI1 to be used as a prognostic marker in gastric, esophageal, nasopharyngeal cancer, prostate, breast, cervical and ovarian cancer, However, the role of BMI1 in maintaining self-renewal and tumorigenicity in HNSCC or HNSCC-derived cancer stem cells (CSCs) remained to be clarified.

ELIGIBILITY:
Inclusion Criteria:

1. In vitro studies.
2. Samples used are oral dysplasia and squamous cell carcinoma.
3. Diagnostic accuracy of Bmi-1 marker on oral dysplasia and SCC.
4. English language published articles only.

Exclusion Criteria:

1. In vivo studies.
2. Studies using any techniques other than immunohistochemistry or PCR.
3. Samples using any carcinoma rather than squamous cell carcinoma.
4. Samples using benign tumors.
5. Samples using sarcomas.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
oral squamous cell carcinoma | 10 months
  Different grades of oral squamous cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Iman A. Radi, Professor, Study Chair — Cairo University
Locations (1):
- Asmaa M. Abou Gabal, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dalley AJ, Pitty LP, Major AG, Abdulmajeed AA, Farah CS. Expression of ABCG2 and Bmi-1 in oral potentially malignant lesions and oral squamous cell carcinoma. Cancer Med. 2014 Apr;3(2):273-83. doi: 10.1002/cam4.182. Epub 2014 Jan 11. PMID 24415717

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT03345966/Prot_SAP_000.pdf